CLINICAL TRIAL: NCT06495424
Title: A Post-Market Observational Multi-Center Study to Evaluate the Effectiveness of Repeated QUTENZA Use in Adults With Painful Diabetic Peripheral Neuropathy of the Feet
Brief Title: Observational Study to Evaluate the Efficacy of Sustained QUTENZA® Use in Painful Diabetic Peripheral Neuropathy
Status: Recruiting | Type: Observational
Sponsor: Averitas Pharma, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AV002
Record Dates: First submitted 2024-07-01; First posted 2024-07-10 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Peripheral Diabetic Neuropathy; Painful Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Capsaicin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study group: All subjects will receive repeat applications of the capsaicin 8% topical system every 12 weeks (up to 3 applications).
  Interventions: Drug: Capsaicin 8%

INTERVENTIONS:
Drug: Capsaicin 8% — Repeat applications every 12 weeks in patients with PDPN of the feet.

SUMMARY:
The purpose of this post-market observational study is to provide real-world evidence to support the repeated use of QUTENZA in patients with PDPN and to evaluate the potential for pain and concomitant medication use reduction.

ELIGIBILITY:
Inclusion Criteria:

1. IRB approved written Informed Consent and privacy language as per national regulations will be obtained from the patient or legally authorized representative prior to any study-related procedures (including withdrawal of prohibited medication, if applicable)
2. Male or female 18 - 80 years of age
3. Diagnosis of painful, distal, symmetrical, sensorimotor polyneuropathy due to diabetes confirmed by the Douleur Neuropathique 4 Interview (DN4I) of at least 3 out of 7
4. Baseline PROMIS-29 numeric pain intensity score over the last 7 days ≥ 4 during the screening period
5. Stable doses of pain medications for PDPN for more than 4 weeks prior to the screening visit
6. Patient agreed not to participate in another interventional study while on treatment

Exclusion Criteria:

1. Pain associated with PDPN in the ankles or above
2. Pain that could not be clearly differentiated from, or conditions that might have interfered with the assessment of the PDPN, such as plantar fasciitis, heel spurs, tibial neuropathy, Morton's neuroma, bunions, metatarsalgia, arthritis in feet, peripheral vascular disease (ischemic pain), neurological disorders unrelated to diabetic neuropathy (eg, phantom limb pain from amputation), skin condition in the area of the neuropathy that could alter sensation (eg, plantar ulcer)
3. Significant pain (moderate or above) of an etiology other than PDPN (eg, compression-related neuropathies [eg, spinal stenosis]), fibromyalgia or arthritis, that may interfere with assessment of PDPN-related pain
4. Current foot ulcer or not intact skin as determined by medical examination
5. Clinically significant foot deformities or foot amputations
6. Any active signs of skin inflammation around onychomycosis sites such as pain, redness, swelling or drainage
7. Patient is unwilling to implement proper foot care methods
8. Diagnosis of any poorly controlled major psychiatric disorder at the Investigator's discretion
9. Evidence of cognitive impairment including dementia that may interfere with patient's ability to complete pain assessments requiring patient's recall of average pain level in the past 24 hours
10. Active substance abuse or history of chronic substance abuse within 1 year prior to screening visit or any prior chronic substance abuse (including alcoholism) likely to have reoccurred during the study period as judged by the Investigator
11. Participation in any other PDPN related clinical study within 30 days prior to the screening visit
12. Previous treatment with QUTENZA
13. Hypersensitivity to capsaicin (eg, chili peppers or over-the-counter capsaicin products) or any QUTENZA excipients
14. Active malignancy or history of malignancy during the past 5 years prior to screening visit (a history of squamous cell carcinoma or a basal cell carcinoma not involving the area to be treated is allowed)
15. Use of transcutaneous nerve or spinal cord stimulators to relieve pain
16. Patient, who in the opinion of the Investigator, is not likely to complete the study for any reason

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients for inclusion in the study are those with PDPN as assessed by the Douleur Neuropathique 4 Interview (DN4I) assessment.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change (%) in pain intensity post QUTENZA administrations | Baseline, weeks 2-12 Post-Admin
  The pain intensity score from baseline will be compared to the average weekly pain intensity score between weeks 2-12 post each QUTENZA application (up to 3 applications).
Change (%) in overall scores for Patient-Report Outcomes Measurement Information System (PROMIS)-29 | Baseline, week 12 Post-Admin
  The baseline PROMIS-29 scores for all domains will be compared to the PROMIS-29 scores assessed at 12 weeks post-each QUTENZA application (up to 3 applications).
Total number of patients who completed each QUTENZA treatment. | week 12 Post-Admin
  Analysis of the number of patients who completed repeated (2 or 3) QUTENZA applications.
Change (%) of concomitant medications at baseline and 12 weeks after each treatment | through study completion, an average of 36 weeks
  The change in utilization of pharmaceutical drug by medication, pharmacology class, dose, and frequency of use for drugs for PDPN, documented by collecting Concomitant medications including indication (for PDPN, for other reasons, and for temporary rescue use for PDPN) and dose

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Pacific Research Institute, Lakeport, California
  - Pacific Research Institute, Santa Rosa, California
  - Pacific Research Institute, Sonoma, California
  - Center for Interventional Pain and Spine, Wilmington, Delaware
  - Horizon Clinical Research, Gainesville, Georgia
  - Horizon Clinical Research, Jasper, Georgia
  - Horizon Clinical Research, Newnan, Georgia
  - Iqra Research, Edgewood, Kentucky
  - Curalta Clinical Trials, Oradell, New Jersey
  - Center for Interventional Pain and Spine, Bryn Mawr, Pennsylvania
  - Center for Interventional Pain and Spine, Fort Washington, Pennsylvania
  - Center for Interventional Pain and Spine, Lancaster, Pennsylvania